CLINICAL TRIAL: NCT01361061
Title: AFP - L3% and DCP as Screening Marker for a Hepatocellular Carcinoma in Patients With Cirrhosis of the Liver- am Multicenter HCC- Surveillance Study
Brief Title: AFP - L3% and DCP as Screening Marker for a Hepatocellular Carcinoma in Patients With Cirrhosis of the Liver
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Collaborators: Wako Diagnostics (Industry); Johannes Gutenberg University Mainz (Other); University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dominik Bettinger, investigator, University Hospital Freiburg
Other Study IDs: HCC3; DRKS00000811 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2011-05-16; First posted 2011-05-26 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2011-12

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; screening; hepatocellular carcinoma; liver cancer markers: AFP, AFP-L3% and DCP
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — measurement of tumor markers AFP, AFP-L3 and DCP in serum samples every 6 months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with liver cirrhosis

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the tumors with a rising incidence worldwide. The aim of this trial is to improve the detection of early HCC nodules in the liver. At the moment screening for HCC in patients with liver cirrhosis is performed by ultrasound and measurement of alpha- fetoprotein (AFP). In this trail the tumor markers AFP- L3 (a subfraction of AFP) and Des-y- carboxyprothromib (DCP) are measured in addition in order to receive information about the course of these markers before the detection of a HCC nodule.

DETAILED DESCRIPTION:
The incidence of the hepatocellular carcinoma (HCC) is rising worldwide. Usually it arises in patients with liver cirrhosis. That's the reason why these patients should be screened every six months by ultrasound performance and by the measurement of alpha-fetoprotein (AFP) in order to detect a growing tumor in the cirrhotic liver so that a possible curative treatment may be possible.

In the last years new tumor markers has been identified such as Des-y- carboxyprothromib (DCP) and AFP - L3. AFP in total consists of three different glycoforms (AFP - L1, AFP - L2 and AFP - L3) which all have a different binding affinity to the lens culinaris agglutinin (LCA). Among these glycoproteins AFP - L3 has the highest binding affinity to LCA and occurs predominantly in patients with a HCC whereas the other subtypes can be found rather in patients with benign diseases of the liver such as a chronic hepatitis or cirrhosis of the liver.

Some studies have shown that high serum levels of AFP - L3 can be associated with a reduced function of the liver, low differentiation and a high malignancy of the HCC. Furthermore HCC - nodules with a diameter smaller than 2 cm could be detected by rising AFP - L3 serum levels. Moreover there are significant differences in AFP - L3 serum levels in patients with cirrhosis of the liver without a HCC and those with such a tumor. In conclusion of that rising AFP - L3 serum levels could indicate a newly developed tumour.

Des-y- carboxyprothromib (DCP), which was first described in 1984 by Liebmann et al. is another tumor marker for HCC. In contrast to AFP it is not elevated in patients with a benign disease of the liver. This could be an interesting fact concerning the screening of patients with liver cirrhosis.

In this examination the diagnostic value of AFP, AFP - L3% and DCP should be evaluated. An important aim of this prospective clinical trial is to define the specificity of these serum markers alone and in combination. If a patient develops a primary liver tumor the course of the tumor markers before the development of the tumor will be analysed. Furthermore it will be examined which parameters will lead to false positive DCP values (especially chronic kidney disease or application of phenprocoumon). During 2 years approximately 150 patients in each center with approved cirrhosis of the liver will be enrolled. According to the normal screening procedure serum samples will be collected for the measurement of AFP, AFP- L3% and DCP. If a suspected tumor nodule is detected, a confirmation of the diagnosis "HCC" according to the AASLD- criteria is needed. These patients will be excluded from the examination and will be treated according to the actual guidelines.

The aim is to improve the early diagnosis of a HCC so that curative treatment opportunities can be done.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80
* cirrhosis of the liver confirmed by ultrasound or other imaging techniques (MRI, CT) or biopsy
* at the time of enrollment: no HCC- suspected lesion detectable in the liver

Exclusion Criteria:

* liver tumors or metastasis or tumor of unknown origin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients approved cirrhosis of the liver, but without a HCC - suspected lesion, are included in this clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2010-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
development of HCC | up to 3 years
  all patients with liver cirrhosis in this clinical trial are examined every 6 months performing ultrasound and measurement of AFP, AFP-L3% and DCP

SECONDARY OUTCOMES:
comparison of these liver cancer markers (AFP, AFP-L3% and DCP) between men and women | baseline
  The levels of these liver cancer markers are compared in men and women and it will be evaluated if one marker is superior than the others in men or women.
comparison of these liver cancer markers (AFP, AFP-L3% and DCP) between different etiologies | baseline
  The levels of these liver cancer markers are compared between different etiologies and it will be evaluated if one marker is superior than the others in different causes of liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Spangenberg, Prof. Dr., Principal Investigator — University Medical Center Freiburg
Locations (2):
- Germany (2):
  - University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Medical Center Mainz, Mainz, Rhineland-Palatinate